CLINICAL TRIAL: NCT00174642
Title: Comparison of Three Therapeutic Strategies for Treating Type 2 Diabetes Mellitus Patients Poorly Controlled With Basal Insulin Associated With Oral Antidiabetic Drugs
Brief Title: Opposing Step-by-step Insulin Reinforcement to Intensified Strategy
Acronym: OSIRIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3506; EUDRACT # : 2004-002036-25
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin glulisine; Metformin

ARMS (3):
- 1 (Experimental): Insulin Glargine + 3 bolus of Insulin Glulisine + Metformin
  Interventions: Drug: Insulin Glargine; Drug: Insulin Glulisine; Drug: Metformin
- 2 (Experimental): Insulin Glargine + 1 to 3 bolus of Insulin Glulisine + Metformin
  Interventions: Drug: Insulin Glargine; Drug: Insulin Glulisine; Drug: Metformin
- 3 (Experimental): Insulin Glargine + 1 to 3 bolus of Insulin Glulisine + Metformin + Insulin secretagogue
  Interventions: Drug: Insulin Glargine; Drug: Insulin Glulisine; Drug: Metformin; Drug: insulin secretagogue

INTERVENTIONS:
Drug: Insulin Glargine — One daily injection in the evening. 100 U/ml
Drug: Insulin Glulisine — Given immediately before each of the three main meals. 100 U/ml
Drug: Metformin — At same dosages as the previous treatment
Drug: insulin secretagogue — sulfonylurea or glinide
  Arms: 3

SUMMARY:
Primary objectives :

* To show the non inferiority in terms of efficacy (HbA1c) of insulin glargine plus metformin combined with 1 to 3 bolus of insulin glulisine introduced progressively (Arm 2) compared with insulin glargine plus metformin combined with 3 bolus of insulin glulisine (Arm 1), in type 2 diabetes mellitus patients poorly controlled on basal insulin therapy with oral antidiabetic drugs.
* To show the non inferiority in terms of efficacy (HbA1c) of insulin glargine plus metformin combined with 1 to 3 bolus of insulin glulisine introduced progressively (Arm 2) compared with insulin glargine plus metformin and insulin secretagogue (sulfonylurea or glinide) combined with 1 to 3 bolus of insulin glulisine introduced progressively (Arm 3), in type 2 diabetes mellitus patients poorly controlled on basal insulin therapy with oral antidiabetic drugs.

Secondary objectives :

* To compare between the 3 treatment groups: evolution of HbA1c over time, percentage of subjects with HbA1c <= 7% at the end of the study, evolution of blood glucose profiles, incidence of hypoglycemia, insulin doses, evolution of body weight and treatment satisfaction.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetic
* BMI ≤ 40 kg/m²
* HbA1c > 7%
* Treated with basal insulin (NPH, Insulin Zinc, insulin glargine or insulin detemir), and at least, two OAD including an insulin secretagogue (sulfonylurea or glinide, at any dosage) and metformin (at the maximum tolerated dosage), for more than 6 months

Exclusion criteria:

* Type 1 diabetes mellitus
* Treatment with OADs only
* Treatment with thiazolidinediones
* Treatment with an insulin other than basal insulin (Premix, rapid insulin, fast-acting insulin analogue)
* Active proliferative diabetic retinopathy, as defined by the application of photocoagulation or surgery, in the 6 months before study entry or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgery during the study (confirmed by an optic fundus performed in the 2 years prior study entry)
* Pregnancy (women of childbearing potential must have a negative pregnancy test at study entry and effective contraception)
* Breast-feeding
* History of hypersensitivity to the study drug or to drugs with a similar chemical structure or to insulin glargine
* Treatment with systemic corticosteroids, irrespective of the dose of administration and irrespective of the prior or foreseeable treatment duration
* Treatment with any investigational product in the last 2 months before study entry, except for insulin glargine
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major disease making implementation of the protocol or interpretation of the study results difficult
* Impaired hepatic function as shown by ALT and/or AST greater than three times the upper limit of normal at study entry
* Impaired renal function as shown by serum creatinine >135 μmol/l in men and > 110 μmol/l in women at study entry
* History of drug or alcohol abuse
* Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* Subject deprived of freedom by a judicial or administrative decision
* Subject is the investigator or any subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2004-12; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | From the beginning to the end of the study
24-hour blood glucose levels | From the beginning to the end of the study
symptomatic hypoglycemia (diurnal and nocturnal) | From the beginning to the end of the study
Severe hypoglycemia (diurnal and nocturnal), | From the beginning to the end of the study
Insulin doses | From the beginning to the end of the study

SECONDARY OUTCOMES:
Vital signs | From the beginning to the end of the study
Adverse events | From the beginning to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, MD, Study Director — Sanofi
Locations (18):
- Sanofi-Aventis, Brussels, Belgium
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Athens, Greece
- Sanofi-Aventis, Budapest, Hungary
- Sanofi-Aventis, Dublin, Ireland
- Sanofi-Aventis, Milan, Italy
- Sanofi-Aventis, Vilnius, Lithuania
- Sanofi-Aventis, México, Mexico
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-Aventis, Moscow, Russia
- Sanofi-Aventis, Seoul, South Korea
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Stockholm, Sweden
- Sanofi-Aventis, Taipei, Taiwan
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis, Guildford, United Kingdom